CLINICAL TRIAL: NCT00707616
Title: The Effect of Diabetes-associated Gene Variation on Glucose Metabolism in Humans
Brief Title: Common Genetic Variation and Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: University of Padova (Other)
Responsible Party: Principal Investigator, Adrian Vella, Professor of Medicine, Mayo Clinic
Other Study IDs: 348-05
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples for hormone measurement and DNA extraction
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Subjects without type 2 diabetes living in Olmsted County, MN
  Interventions: Other: Oral glucose tolerance test

INTERVENTIONS:
Other: Oral glucose tolerance test — one time 75g oral glucose tolerance test for measurement of insulin secretion and action

SUMMARY:
Type 2 diabetes is a common metabolic disorder arising from a complex interaction between genetic predisposition and the environment. The development of this disorder is preceded by impaired glucose tolerance and elevated fasting glucose which also carry adverse cardiovascular risk. To date a few common genetic variants have been reliably associated with predisposition to type 2 diabetes. However, it is uncertain how these genes interact to alter insulin secretion and insulin action prior to the development of type 2 diabetes. We propose to utilize an established population-based cohort to determine how common genetic variants associated with type 2 diabetes alter the response to an oral glucose challenge in people without overt type 2 diabetes. This will enable us to understand how common variants alone or in combination alter whole-body glucose physiology and predispose to type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Fasting blood glucose < 126mg/dL

Exclusion Criteria:

* Fasting blood glucose > 126mg/dL

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy, non-diabetic
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2006-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Disposition Index | 2 hr
  Measured by 7-sample, 2Hr OGTT

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States